CLINICAL TRIAL: NCT06727331
Title: Tirzepatide for the Treatment of Alcohol Use Disorder: A Pilot Randomized Controlled Trial
Brief Title: Study of Tirzepatide for Recovery and Alcohol Use Management
Acronym: STREAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024P003497
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The IDS will perform both the randomization and blinding and will be the only unblinded research staff. They will extract the tirzepatide and draw the dose into syringes, which will match visually with the placebo doses. All other research staff will remain blinded for the duration of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide (Experimental): This arm will receive tirzepatide (n=10) weekly 2.5mg injections for 4 weeks.
  Interventions: Drug: Tirzepatide
- Saline Placebo (Placebo Comparator): This arm will receive saline placebo injections (n=10) weekly for 4 weeks.
  Interventions: Other: Saline Placebo

INTERVENTIONS:
Drug: Tirzepatide — This intervention will consist of the FDA-approved dosing schedule. Participants will receive 2.5mg weekly injections for 4 weeks. IDS will extract tirzepatide and draw the doses into syringes.
  Other Names: Mounjaro
  Arms: Tirzepatide
Other: Saline Placebo — Placebo syringes of saline and matching volume will be produced by IDS.
  Arms: Saline Placebo

SUMMARY:
This is a pilot, 4-week, double-blind, placebo-controlled, randomized trial of individuals with alcohol use disorder (AUD) to receive weekly injections of either tirzepatide (n=10) or matching placebo (n=10). The primary aim is to determine the effects of tirzepatide on cue-reactivity among individuals with AUD. The secondary aim is to assess the safety and preliminary efficacy of tirzepatide for AUD.

DETAILED DESCRIPTION:
Participants include N=20 men and women with DSM5 diagnosis of AUD. Potential participants will be screened and enrolled only if they meet full inclusion criteria. After screening and baseline procedures (Visit 1) are complete, participants will be randomized to receive either tirzepatide or placebo. Following randomization, participants will be scheduled for five study visits (Visits 2-6). Each visit will last approximately 1 hour, except for study visits 1 and 6 which will take no more than 3 hours in order to conduct additional neurocognitive testing, including cue-induced cravings and decision-making tests. At all study visits, participants will complete vital signs, weight, urine toxicology testing, a blood draw for glucose, and questionnaires probing secondary outcomes (i.e. anxiety and depression, suicidality, substance use, opioid withdrawal symptoms, cravings, etc). At study visits 2-5, the weekly dose of tirzepatide or placebo will be administered, and assessment of adverse events will also be completed. Both participants and study staff (including raters) will be blinded to active drug vs. placebo. At visit 1, subjects' expectations about their potential treatment will be queried. The final visit, visit 6, also called the follow-up visit, will also assess subjects' guess as to which treatment they received. The medication will be purchased from the manufacturer and stored by IDS. The IDS will extract the tirzepatide and draw the dose into syringes, which will match visually with the placebo doses.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults aged 18 and above
* Diagnosed with current DSM-5 alcohol use disorder
* Willing and able to physically travel to BWH CCI outpatient facilities for study visits

Exclusion Criteria:

* CIWA score at screening ≥ 8.
* Psychotic disorder, active suicidality or homicidality or any psychiatric condition that impair ability to provide informed consent
* Any lifetime diagnosis of eating disorders including anorexia, bulimia, binge eating, or avoidant/restrictive food intake disorder
* BMI<23 mg/kg2
* Current or lifetime diagnosis of Type 1 or Type 2 diabetes
* Current (or within 30 days of enrollment) use of any anti-obesity medications or medications with glucose lowering properties (including GLP-1 analogues, sulfonylurea, insulin, metformin, thiazolidinediones, dipeptidyl peptidase-4 (DPP-IV) inhibitors, or sodium-glucose cotransporter-2 (SGLT-2) inhibitors)
* Use of any GLP-1 agonist medications in the prior 3 months
* Anticipating receipt of any other GLP-1 agonist medications during the trial
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Current hypoglycemia as indicated by a blood sugar level of ≤70 mg/dL measured at the baseline visit
* Calcitonin ≥ 50 ng/L
* Triglycerides ≥500 mg/dL
* Untreated cholelithiasis or gallbladder disease
* Acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, or congestive heart failure in the last 90 days
* Uncontrolled hypertension at baseline, as indicated by an average blood pressure reading of >180/110 after three successive readings
* History of inflammatory bowel disease, bariatric surgery, pancreatitis, diabetic gastroparesis, or non-arteritic anterior ischemic optic neuropathy
* Liver function test greater than 5 times upper normal limit
* Renal impairment as indicated by eGFR of <30
* History of hypersensitivity or allergy to tirzepatide
* Pregnant or breastfeeding
* Anticipated to be enrolled in another clinical drug trial during participation in this trial
* Any other reason or clinical condition that the investigators judge may interfere with study participation and/or be unsafe for a participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cue-induced Cravings for Alcohol | Baseline visit and 5 weeks after baseline visit.
  Cue-induced craving scores at follow-up compared to baseline using a standard cue-reactivity paradigm utilizing visual cues. Cravings will be measured on a scale from 0-10 with 10 meaning extreme cravings.
Incidence and Severity of Adverse Events | Epic monitoring throughout the trial and PRISE administered at study weeks 2-5 (visits 3-6).
  Study staff will be notified of any hospital admissions via Epic, and adverse events will be queried specifically using the Patient Rated Inventory of Side Effects (PRISE) at study weeks 2-5. The PRISE is a self-report tool to qualify side effects. For each domain, the patient indicates whether they have experienced certain symptoms and whether the symptoms are tolerable or distressing.

SECONDARY OUTCOMES:
Penn Alcohol Craving Scale (PACS) | At each study visit up to and including the final visit 5 weeks after baseline.
  A self-report tool used to measure craving for alcohol during the past week. Participants respond to 5 questions on a scale of 0-6 for a total score of 0-30, with higher scores indicating stronger cravings.
Monetary Choice Questionnaire (MCQ) | Baseline visit and 5 weeks after baseline visit.
  A self-report tool used to measure delayed discounting. Participants will be asked to pick one of the two choices given. Score calculated typically falls between 0.0 and 0.5, with smaller values indicating a lack of discounting and preference for delayed rewards and higher values indicating strong discounting and a preference for immediate rewards.
Visual Probe Task | Baseline visit and 5 weeks after baseline visit.
  A behavioral task to assess attentional bias. Alcohol-related and neutral images will be used, different from the ones used for the cue-reactivity paradigm to limit habituation. A pair of images will appear on the left and right of the screen for either a short (200ms) or long (500ms) stimulus duration to assess automatic orientating and controlled attention processing, respectively. Image pairs will be replaced by a probe in the location of either the opioid-related or neutral image. The probe will remain until the participant responds to identify the probe orientation by pressing the response keys as quickly as possible. This task will yield reaction times for analysis.
Percent days abstinent | At each study visit up to and including the final visit 5 weeks after baseline.
  The percentage of days abstinent from alcohol, defined as 0 drinks on a given day, out of all days queried. The study investigators will use the Time-Line Follow Back (TLFB), a gold-standard method of evaluating substance use, as well as weekly urine toxicology screens.
Percent heavy drinking days | At each study visit up to and including the final visit 5 weeks after baseline.
  Percentage of heavy drinking days, defined as 5 or more drinks in one day for males and 4 or more drinks in one day for females, out of all days queried. The study investigators will use the Time-Line Follow Back (TLFB), a gold-standard method of evaluating substance use, as well as weekly urine toxicology screens.
Drinks per drinking day | At each study visit up to and including the final visit 5 weeks after baseline.
  The average number of drinks per drinking day. A drinking day is a day in which one or more alcoholic beverages were consumed. The study investigators will use the Time-Line Follow Back (TLFB), a gold-standard method of evaluating substance use, as well as weekly urine toxicology screens.
Clinical Institute Withdrawal Assessment (CIWA) | At each study visit up to and including the final visit 5 weeks after baseline.
  Tool for assessing alcohol withdrawal. Scale of 0-67, with a higher number meaning more severe withdrawal.
Blood Sugar | At each study visit up to and including the final visit 5 weeks after baseline.
  Blood glucose obtained via finger stick or blood already drawn for other tests.
Hemoglobin A1c | Baseline and 5 weeks after baseline visit.
  Hemoglobin A1c obtained via blood draw.
Weight | At each study visit up to and including the final visit 5 weeks after baseline.
  Weight measured in kilograms.
Columbia Suicide Severity Rating Scale (C-SSRS) | At each study visit up to and including the final visit 5 weeks after baseline.
  A commonly used tool to assess suicidal ideation. The sum ranges from 2 to 25, with the higher number indicating more intense ideation.
Patient Health Questionnaire-8 (PHQ-8) | At each study visit up to and including the final visit 5 weeks after baseline.
  A tool to assess depression symptoms. Scale of 0-24, with a higher score meaning more depression symptoms.
Generalized Anxiety Disorder-7 (GAD-7) | At each study visit up to and including the final visit 5 weeks after baseline.
  A standard tool to assess anxiety symptoms. Scale of 0-21 with a higher number indicating more anxiety.
Heart rate | At each study visit up to and including the final visit 5 weeks after baseline.
  Heart rate measured in beats per minute.
Blood pressure | At each study visit up to and including the final visit 5 weeks after baseline.
  Blood pressure measured in systolic/diastolic (mmHg/mmHg). mmHg = millimeters of mercury.
Assessment of Blind | 5 weeks after baseline visit.
  Measure of participant perception of whether they received the active study drug.
Stanford Efficacy of Treatment Scale (SETS) | Baseline visit.
  A tool for measuring patient outcome expectancy in clinical trials.
Fibrosis-4 (FIB-4) | Baseline visit and 5 weeks after baseline visit.
  A non-invasive measure of liver fibrosis. The higher the score, the more severe the fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Joji Suzuki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Jamaica Plain, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided